CLINICAL TRIAL: NCT07138092
Title: Comparison of Gastric Insufflation Volume by Ultrasound Using I-gel and ProSeal Laryngeal Mask Airways in Patients Undergoing Urological Surgery
Brief Title: Comparison of Gastric Volume in I-gel and ProSeal Laryngeal Mask Airways
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Diskapi Yildirim Beyazit Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Zeynep Koc, principal investigator, Diskapi Yildirim Beyazit Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZeynepKoc006
Record Dates: First submitted 2025-08-15; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Nausea and Vomiting, Postoperative; Sore-throat
Keywords: Gastric insufflation; Ultrasound; Supraglottic airway devices; Oropharyngeal leak pressure
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Pharyngitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- i jel group (Experimental): under general anesthesia, patients inserted i jel LMA
  Interventions: Other: i jel LMA
- proseal group (Experimental): under general anesthesia, patients inserted proseal LMA.
  Interventions: Other: proseal LMA

INTERVENTIONS:
Other: i jel LMA — Patients will be inserted i jel laryngeal mask under general anesthesia.
  Arms: i jel group
Other: proseal LMA — Patients will be inserted proseal laryngeal mask under general anesthesia.
  Arms: proseal group

SUMMARY:
This study was planned to compare the gastric insufflation volume between i jel and ProSeal laryngeal mask airway (LMA) and its relationship with the oropharyngeal sealing pressure and the incidence of postoperative complications in patients undergoing urological surgery.

DETAILED DESCRIPTION:
Supraglottic airway devices (SADs) are widely used in both elective and emergency surgeries, resuscitation, and difficult airway management. Compared to endotracheal intubation, they are less invasive, require lower doses of anaesthetic agents, and cause less haemodynamic instability. Among supraglottic airway devices, the I-gel differs from other SADs in that it does not have an inflatable cuff; instead, it features a soft structure made of a transparent thermoplastic elastomer that mimics a cuff. In addition, it has a gastric channel alongside the airway tube that allows for gastric aspiration.

ProSeal LMA is one of the most commonly used SADs in clinical practice. It was developed in the early 2000s as a modification of the classic LMA and includes an inflatable cuff. Like the I-gel, it also features a gastric drainage channel for aspiration.

Aspiration pneumonia is a serious complication of anaesthesia, accounting for approximately 9% of all anaesthesia-related mortality. Traditionally, oropharyngeal leak pressure (OLP) provides information about the potential for gastric insufflation and thus the risk of gastric aspiration. Measurement of the gastric antral cross-sectional area (AGCA) by ultrasound allows for the estimation of gastric volume and helps assess the risk of aspiration.

This study was planned to compare the gastric insufflation volume between i jel and ProSeal LMA and its relationship with the oropharyngeal sealing pressure and the incidence of postoperative complications in patients undergoing urological surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an ASA (American Society of Anesthesiologists) physical status score of 1 to 3
* undergoing urological surgeries performed with I-gel or ProSeal LMA

Exclusion Criteria:

* Difficult airway
* Clinically significant upper respiratory tract infection
* Pre-existing airway disease
* Pre-existing airway disease
* History of head and neck surgery
* Pregnant patients
* Patients with upper gastrointestinal tract disease

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-08-18 (Estimated); Primary Completion 2025-09-29 (Estimated); Study Completion 2025-10-10 (Estimated)

PRIMARY OUTCOMES:
Measurement of oropharyngeal leak pressure (OLP) | Five minutes after successful LMA placement
  One minute after successful LMA placement and fixation, oropharyngeal leak pressure (OLP) will be measured by setting the adjustable pressure limiting valve (APL) to 40 mmHg and maintaining a fresh gas flow of 3 L/min. The OLP will be recorded as the pressure at which an audible leak sound is heard from the mouth.

SECONDARY OUTCOMES:
Gastric volume | 1 minute before induction of anesthesia
  Before induction of anesthesia, gastric ultrasonography will be performed by an experienced anaesthesiologist using a 2-5 MHz curved-array probe. The gastric antrum will be visualised in the sagittal plane in the epigastric region, located between the left lobe of the liver anteriorly, the aorta or inferior vena cava inferiorly, and the pancreas posteriorly.
  The gastric cross-sectional area (CSA) will be calculated using the following formula, assuming the antrum is elliptical: CSA = (A × B × π) / 4, where A is the anteroposterior diameter and B is the craniocaudal diameter. The estimated gastric volume will be calculated using a previously validated model for non-pregnant adults: Estimated gastric volume (mL) = 27 + (14.6 × ACSA [cm²]) - (1.28 × Age [years]).
Gastric volume | End of the operation, 5 minutes before LMA removal,
  End of the operation,befeore LMA removal gastric ultrasonography will be performed by an experienced anaesthesiologist using a 2-5 MHz curved-array probe. The gastric antrum will be visualised in the sagittal plane in the epigastric region, located between the left lobe of the liver anteriorly, the aorta or inferior vena cava inferiorly, and the pancreas posteriorly.
  The gastric cross-sectional area (CSA) will be calculated using the following formula, assuming the antrum is elliptical: CSA = (A × B × π) / 4, where A is the anteroposterior diameter and B is the craniocaudal diameter. The estimated gastric volume will be calculated using a previously validated model for non-pregnant adults: Estimated gastric volume (mL) = 27 + (14.6 × ACSA [cm²]) - (1.28 × Age [years]).
fiberoptic view grading | Five minutes after successful LMA placement
  The Brimacombe score will be used to evaluate the view obtained with fiberoptic bronchoscopy. 1: Vocal cords are not visible; 2: Vocal cords and anterior epiglottis are visible; 3: Vocal cords and posterior epiglottis are visible; 4: Vocal cords are visible.
Complications during i jel and propseal LMA removal (emerge) | One minute after i jel and propseal LMA removal
  Complications during SP_Air-Q and proseal LMA removal (emerge) such as breath-holding during emergence, airway obstruction, coughing, hypoxia (SpO2 < 90%), vomiting, lip-tongue-teeth trauma, and bleeding, will be recorded.

OTHER OUTCOMES:
sore throat | popstoperative 1. hour
  The presence or absence of sore throat will be recorded at the firsth postoperative hour.
sore throat | popstoperative 24. hours
  The presence or absence of sore throat will be recorded at the firsth postoperative hour.
dysphonia | popstoperative 1. hour
  The presence or absence of dysphonia will be recorded at the firsth postoperative hour.
dysphonia | 24 hours postoperatively
  The presence or absence of dysphonia will be recorded at the 24th postoperative hour.

CONTACTS AND LOCATIONS:
Locations (1):
- Zeynep Koç, Yenimahalle, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gunasekaran A, Govindaraj K, Gupta SL, Vinayagam S, Mishra SK. Comparison of Gastric Insufflation Volume Between Ambu AuraGain and ProSeal Laryngeal Mask Airway Using Ultrasonography in Patients Undergoing General Anesthesia: A Randomized Controlled Trial. Cureus. 2022 Aug 11;14(8):e27888. doi: 10.7759/cureus.27888. eCollection 2022 Aug. PMID 36110490
- [Background] Zhou S, Cao X, Zhou Y, Xu Z, Liu Z. Ultrasound Assessment of Gastric Volume in Parturients After High-Flow Nasal Oxygen Therapy. Anesth Analg. 2023 Jul 1;137(1):176-181. doi: 10.1213/ANE.0000000000006340. Epub 2023 Jan 11. PMID 36630297
- [Result] Ye Q, Wu D, Fang W, Wong GTC, Lu Y. Comparison of gastric insufflation using LMA-supreme and I-gel versus tracheal intubation in laparoscopic gynecological surgery by ultrasound: a randomized observational trial. BMC Anesthesiol. 2020 Jun 3;20(1):136. doi: 10.1186/s12871-020-01057-z. PMID 32493213